CLINICAL TRIAL: NCT02545036
Title: Clinical Study of Combined Western Medicine and Traditional Chinese Medicine Daycare Model for Chronic Kidney Disease Patients
Brief Title: Combined Western and Traditional Chinese Medicine Daycare for CKD Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Collaborators: Ministry of Health and Welfare, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMUH104-REC1-041
Record Dates: First submitted 2015-06-25; First posted 2015-09-09 (Estimated); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Chronic Kidney Disease
Keywords: chronic kidney disease; Daycare; Traditional Chinese Medicine(TCM)
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Medicine, Chinese Traditional

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TCM daycare model (Experimental): 30 patients will be assigned to this arm. The assignment depends on the patients' own will. After diagnosis by nephrology physician, these patients will be distributed to control group by their wills. The intervention is Traditional Chinese Medicine (TCM) daycare model, which provides multiple approaches of traditional Chinese medical treatment, including 5 tones of Chinese music, massage on meridians and collaterals, acupuncture, and patient education. The treatment course is one time a week, for 12 weeks (12 treatments in total). And the model will be provided by a team work clinical care system organized by doctors, nurses, pharmacists and case managers, also provide a comprehensive TCM care system for every visit.
  Interventions: Other: Traditional Chinese Medicine (TCM) daycare model
- Control group (No Intervention): 30 patients will be assigned to this arm. The assignment depends on the patients' own will. After diagnosis by nephrology physician, these patients will be distributed to control group by their wills. The control group will only receive assessment and follow-up without intervention.

INTERVENTIONS:
Other: Traditional Chinese Medicine (TCM) daycare model — Traditional Chinese Medical (TCM) daycare model provides multiple approaches of traditional Chinese medical treatment, including 5 tones of Chinese music, massage for meridians and collaterals, acupuncture, and patient education. The treatment course is one time a week, for 12 weeks (12 treatments in total).
  Arms: TCM daycare model

SUMMARY:
The annual report of USRDS shows than Taiwan has the highest prevalence of end-stage-renal-disease globally resulted in high prevalence dialysis rate. The major factors associated with chronic renal failure are age, diabetes, hypertension, chronic glomerulonephritis, metabolic syndrome, smoke, hepatitis C, painkiller and herbals. Chronic kidney disease may lead to various metabolic, cardiovascular and neurological diseases. And these possible prognostic factors associating with the disease progression and ultimately increase the morbidity and mortality. End-stage renal failure is an irreversible course often with clinical manifestations of edema, fatigue, anemia and uremic pruritus. Patients often use Chinese medicine or acupuncture to help them to ease the symptom.

The aim of this study is to investigate the efficacy of combined Western medicine and traditional Chinese medicine daycare model for chronic kidney disease patients. The study approach to investigate whether combination of Western medicine and traditional Chinese medicine daycare model can improve the clinical symptoms and quality of life as well as the laboratory biochemistries data.

DETAILED DESCRIPTION:
Keywords：chronic kidney disease , Day care, Traditional Chinese Medicine(TCM)

Background and purpose:

The annual report of USRDS shows than Taiwan has the highest prevalence of end-stage-renal-disease globally resulted in high prevalence dialysis rate. The major factors associated with chronic renal failure are age, diabetes, hypertension, chronic glomerulonephritis, metabolic syndrome, smoke, hepatitis C, painkiller and herbals. Chronic kidney disease may lead to various metabolic, cardiovascular and neurological diseases. And these possible prognostic factors associating with the disease progression and ultimately increase the morbidity and mortality. End-stage renal failure is an irreversible course often with clinical manifestations of edema, fatigue, anemia and uremic pruritus. Patients often use Chinese medicine or acupuncture to help them to ease the symptom.

The aim of this study is to investigate the efficacy of combined Western medicine and traditional Chinese medicine daycare model for chronic kidney disease patients. The study approach to investigate whether combination of Western medicine and traditional Chinese medicine daycare model can improve the clinical symptoms and quality of life as well as the laboratory biochemistries data.

Material and methods:

A total of 60 volunteers of patients with chronic kidney disease will be recruited from the Chinese medicine or Western medicine clinics. After diagnosis by nephrology physician, 30 patients will be distributed to combinational Western and TCM daycare model, one time a week, for 12 weeks (12 treatment in total). Another 30 patients will enter Western daycare model. The assignment depends on the patients' own will. The TCM day care model will be provided by a team work clinical care system organized by doctors, nurses, pharmacists and case managers. This model will provide a comprehensive TCM care system for every visit. Laboratory biochemistries analysis and other questionnaires including SF36 health survey, Pittsburgh Sleep Quality Index, Beck Depression Inventory-II, FACIT-fatigue Scale and the 5-D itch scale will be completed at baseline, 6weeks, and 12 weeks after join this study. Instrumental examinations including heart rate variability and traditional Chinese medicine four examinations will be given before and after intervention.

Predict results:

The investigators expect that the efficacy of this combined western medicine and traditional Chinese medicine day care model will be superior to the "pre-ESRD prevention and education program" which execute since 2006 in improving edema, fatigue, physical function and quality of life. The effectiveness of combined therapy can be measured by questionnaires. Moreover, the investigators will further speculate the mechanism by analyzing laboratory data.

ELIGIBILITY:
Inclusion Criteria:

1. Fit CKD definition by National Kidney Foundation's Kidney Disease Outcome Quality Initiative（NKF-KDOQI, pre-ESRD stage IIIb~IV (GFR: 15-44).
2. at least 20 years old volunteers.
3. The participants had no allergy to acupuncture needle in the past, or without contraindications to acupuncture treatment.
4. The participants agreed to join the trial and sign informed consent form after thorough explanation.

Exclusion Criteria:

1. Age less than 20 years old.
2. Using immunosuppressive drug or receiving chemotherapy.
3. Had substance abuse in the past, or having substance abuse.
4. Pregnancy women or breastfeeding women.
5. Mental or behavioral disorders which leads to inability to cooperation.
6. Arrhythmia patients who have pacemaker.
7. Patient who have skin infection or wound infection near acupoints.
8. Patient who have coagulation abnormalities or low platelet count by blood tests (platelet≤150000 / uL).
9. Participating other clinical trials.
10. Patient with serious diseases such as myocardial infarction, severe arrhythmia, heart failure, chronic obstructive airway disease, or cancer.
11. Patients who have limb edema and severe skin lesions not suitable for acupuncture or massage.
12. Patients who took Chinese herbal medicine or received acupuncture treatment in the past 2 weeks.
13. Patients who disagree to sign informed consent form.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2015-06; Primary Completion 2016-11-01 (Actual); Study Completion 2017-09-20 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Creatinine(mg/dL) at 3 months | baseline,12th week
Change from Baseline in GFR(ml/min/1.73m2)at 3 months | baseline,12th week

SECONDARY OUTCOMES:
The Pittsburgh Sleep Quality Index | baseline, 6th ,12th week
Beck Depression Inventory II | baseline, 6th ,12th week
FACIT-fatigue scale | baseline, 6th ,12th week
The 5-D itch scale | baseline, 6th ,12th week
skin pruritus on Visual Analogue Scale | baseline, 6th ,12th week
  for skin pruritus
TCM body constitution questionnaire | baseline, 6th ,12th week
heart rate variability | baseline, 12th week
TCM diagnosis | baseline, 12th week
SF-36 Health Survey | baseline, 6th ,12th week

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, Taiwan